CLINICAL TRIAL: NCT03598296
Title: Comparison of the Results of Two Chest Tube Management During an Enhanced Recovery Program After Video-Assisted Thoracoscopic Lobectomy.
Brief Title: The Affection of Two Chest Management for Enhanced Recovery Program After Video-assisted Thoracoscopic Lobectomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201805
Record Dates: First submitted 2018-06-07; First posted 2018-07-26 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Chest Tube
Keywords: ERAS(Enhanced Recovery After Surgery); Video-assisted thoracoscope lobectomy; Non-Small Cell Lung Cancer (NSCLC); Chest tube
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Total 60 patients accept video-Assisted thoracoscopic lobectomy are divided into two groups(Group A and Group B) equally and randomly.Different group takes different chest tube managements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A:Group Tube (Experimental): Patients are inserted the large size tube (28F).Patients undergo upper lobectomy are inserted one additional large size tube(28F,we named this tube upper tube).This group is planned to enroll 30 patients.
  Interventions: Other: Large size tube
- Group B:Group Ball (Experimental): Patients are inserted the small size tube connects with a negative pressure ball(drainage ball).Patients undergo upper lobectomy are inserted one additional large size tube(28F,we named this tube upper tube).This group is planned to enroll 30 patients.
  Interventions: Other: Drainage ball

INTERVENTIONS:
Other: Large size tube — Patients in Group A are inserted the large size tube (28F).
  Other Names: Upper tube
  Arms: Group A:Group Tube
Other: Drainage ball — Patients in Group B are inserted the small-bore tube connects with a negative pressure ball(drainage ball).
  Other Names: Upper tube
  Arms: Group B:Group Ball

SUMMARY:
Comparing the influences of different chest tube managements for enhanced recovery program after video-Assisted thoracoscopic lobectomy.

DETAILED DESCRIPTION:
The Enhanced Recovery Program has a series of observation data contains hospitalization days, adverse events, drainage, extubation, visual analogue scale(VAS) scores and the number of analgesic using.The investigators plan to enroll 60 patients and divide them into two groups to compare the influences of different chest tube managements for enhanced recovery program after video-assisted thoracoscopic lobectomy.

ELIGIBILITY:
Inclusion Criteria:

* Only single lesion on the targeted lobe
* Considered as invasive carcinoma by preoperative computed tomography (CT) or -diagnosed by intraoperative pathology
* Patients have signed informed consent.

Exclusion Criteria:

* Patients have critical basic disease(diabetes and hypertension).
* Patients who lung function cannot undertake the lobectomy.
* The lesion has the possibility of metastasis.
* Finding serious adhesion to pleura during operation

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-28 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-10-27 (Actual)

PRIMARY OUTCOMES:
Hospitalization days | From the first days after surgery to discharge,up to 4 weeks.
  The numbers of days of patients stay in the hospital after surgery

SECONDARY OUTCOMES:
VAS scores | Pain is measured by VAS on the first 24 hours of after operation and the first 24 hours after tube removing.
  VAS(Visual Analogue Score) is a method to value the degree of patient's pain after surgery.This method has a scale range from 1 to 10.Patient chose a number from it to represent his(her) pain.The "1" represents painless and the "10" represents sever pain which he(she) unable to bear. The pain is increasing with the increasing of number.
Analgesics | Counting the total analgesics using times through study completion, an average of 3 months.
  The number of analgesics using after surgery.
Drainage | Measure the volume every 24 hours,up to 4 weeks
  The total volume of fluid.
Pulmonary recruitment | The first 24 hours after surgery and 8 hours before leaving hospital.
  Chest X-Ray
Adverse event | Counting the times of adverse events through study completion, an average of 3 months.
  Air-leakage or seepage from the surrounding of tube.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Jun, Study Director — The First Affiliated Hospital of Soochow University; Cui zihan, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- First Affiliated Hospital, Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wisely JC, Barclay KL. Effects of an Enhanced Recovery After Surgery programme on emergency surgical patients. ANZ J Surg. 2016 Nov;86(11):883-888. doi: 10.1111/ans.13465. Epub 2016 Mar 17. PMID 26990499
- [Result] Ettinger DS, Wood DE, Aisner DL, Akerley W, Bauman J, Chirieac LR, D'Amico TA, DeCamp MM, Dilling TJ, Dobelbower M, Doebele RC, Govindan R, Gubens MA, Hennon M, Horn L, Komaki R, Lackner RP, Lanuti M, Leal TA, Leisch LJ, Lilenbaum R, Lin J, Loo BW Jr, Martins R, Otterson GA, Reckamp K, Riely GJ, Schild SE, Shapiro TA, Stevenson J, Swanson SJ, Tauer K, Yang SC, Gregory K, Hughes M. Non-Small Cell Lung Cancer, Version 5.2017, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2017 Apr;15(4):504-535. doi: 10.6004/jnccn.2017.0050. PMID 28404761
- [Result] Bertolaccini L, Rocco G, Crisci R, Solli P. Enhanced recovery after surgery protocols in video-assisted thoracic surgery lobectomies: the best is yet still to come? J Thorac Dis. 2018 Mar;10(Suppl 4):S493-S496. doi: 10.21037/jtd.2018.02.33. No abstract available. PMID 29629194
- [Result] Gottgens KW, Siebenga J, Belgers EH, van Huijstee PJ, Bollen EC. Early removal of the chest tube after complete video-assisted thoracoscopic lobectomies. Eur J Cardiothorac Surg. 2011 Apr;39(4):575-8. doi: 10.1016/j.ejcts.2010.08.002. Epub 2010 Sep 15. PMID 20833554
- [Result] Xie HY, Xu K, Tang JX, Bian W, Ma HT, Zhao J, Ni B. A prospective randomized, controlled trial deems a drainage of 300 ml/day safe before removal of the last chest drain after video-assisted thoracoscopic surgery lobectomy. Interact Cardiovasc Thorac Surg. 2015 Aug;21(2):200-5. doi: 10.1093/icvts/ivv115. Epub 2015 May 15. PMID 25979532
- [Derived] Cui Z, Zhang Y, Xu C, Ding C, Chen J, Li C, Zhao J. Comparison of the results of two chest tube managements during an enhanced recovery program after video-assisted thoracoscopic lobectomy: A randomized trial. Thorac Cancer. 2019 Oct;10(10):1993-1999. doi: 10.1111/1759-7714.13183. Epub 2019 Sep 2. PMID 31475791